CLINICAL TRIAL: NCT01094990
Title: Efficacy of Dexamethasone for The Prevention of Nausea and Vomiting Associated With Intrathecal Chemotherapy and Ketamine Sedation in Children With Leukemia
Brief Title: Efficacy of Dexamethasone for Prevent Vomiting in Leukemic Children Who Receive Intrathecal Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CHANCHAI TRAIVAREE (Other)
Responsible Party: Sponsor-Investigator, CHANCHAI TRAIVAREE, Phramongkutklao College of Medicine and Hospital, Phramongkutklao College of Medicine and Hospital
Organization: Phramongkutklao College of Medicine and Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DEX111; PMK111 (Other: Pharmongkutklao)
Record Dates: First submitted 2010-03-26; First posted 2010-03-29 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Acute Leukemic Patients in Children
Keywords: crossover; double blinded; intrathecal chemotherapy; dexamethasone; ketamine;vomiting
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Dexamethasone — dexamethasone 0.25 mg/kg (8 mg/m2/dose) intravenous one time

SUMMARY:
Null hypothesis The proportions of vomiting are not different between dexamethasone and placebo in the patient after sedation with intravenous ketamine and lumbar puncture with intrathecal chemotherapy Alternative hypothesis The proportions of vomiting are different between dexamethasone and placebo in the patient after sedation with intravenous ketamine and lumbar puncture with intrathecal chemotherapy

DETAILED DESCRIPTION:
Does intravenous dexamethasone 0.25 mg/kg (8 mg/m2/dose) have an effect in the reduction of vomiting and retching after sedation with intravenous ketamine and lumbar puncture with intrathecal chemotherapy comparison with placebo?

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 2-15 years who underlying acute lymphoid or nonlymphoid leukemia and need to receive ketamine and intrathecal chemotherapy.
* Personally signed and dated informed consent and assent document indicating that the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to study entry.

Exclusion Criteria:

* Patients who had a known allergy to ketamine or dexamethasone.
* Patients who had contraindication for ketamine or dexemethasone such as hypertension, increased intracranial pressure or central nervous system mass lesion, major psychiatric , and hyperglycemia.
* Patients who concurrent with nausea and vomiting during that time.
* Patients who received ondansetron or other antiemetic before doing Procedure.
* Patients who received other chemotherapy before or after 24 hours.

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
: To determine whether vomiting and retching associated with intravenous ketamine and intrathecal chemotherapy may be reduced by the addition of prophylactic dexamethasone | 24 hours

SECONDARY OUTCOMES:
To determine whether severity of the nausea after procedure may be reduced by the addition of prophylactic dexamethasone. | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: chanchai traivaree, MD, Principal Investigator — Phramongkutklao College of Medicine and Hospital
Locations (2):
- Thailand (2):
  - Phramongkutklao hospital, Bangkok, Bangkok
  - Phramongkutklao Hospital, Bangkok, Bangkok